CLINICAL TRIAL: NCT05284162
Title: Effects of a Theory-guided Health Coaching Programme on Health Promoting Behaviours in Middle-Aged Adults With Cardiometabolic Risk: a Randomised Controlled Trial
Brief Title: Health Coaching Programme on Health Promoting Behaviours in Middle-Aged Adults With Cardiometabolic Risk
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Zoe Ching Man Kwok, Principal Investigator, Lecturer, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Health coaching midlife CMD
Record Dates: First submitted 2022-02-27; First posted 2022-03-17 (Actual); Last update posted 2022-03-17 (Actual); Status verified 2022-03

CONDITIONS: Coaching; Cardiovascular Diseases; Metabolic Diseases
Keywords: Health coaching; Health promoting behaviour; Cardiometabolic disease; Middle-aged
MeSH Terms: conditions — Cardiovascular Diseases; Metabolic Diseases; Health Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Health coaching (Experimental): Health coaching
  Interventions: Behavioral: Health coaching
- Usual care (No Intervention): Usual care

INTERVENTIONS:
Behavioral: Health coaching — The health coaching program includes four monthly health coaching sessions for three months.
  Arms: Health coaching

SUMMARY:
Cardiometabolic disease has been an increasing trend globally and remains the major cause of morbidity and mortality in Hong Kong. Health coaching intervention are generally effective for managing chronic disease and prevention of complication. However, there is fewer attention on the effects of health coaching in primary disease prevention. This study aims to evaluate the effects of health coaching programme on increasing health promoting behaviours in middle-aged adults with cardiometabolic risk.

DETAILED DESCRIPTION:
Cardiometabolic disease, including metabolic syndrome, prediabetes, type 2 diabetes mellitus, coronary heart disease, myocardial infarction and stroke, has been an increasing trend globally, and increased more than double over 5 years in China [1].

Cardiometabolic disease remains the major cause of morbidity and mortality in Hong Kong [2]. Type 2 diabetes mellitus is associated with increased risk for morbidity and mortality [3]. Ischaemic heart disease and stroke were the major cause of disability-adjusted life years (DALYs) worldwide, resulting in dependence, disability and cognitive impairment [4]. Moreover, midlife stroke risk is associated with cognitive decline within 10 years [5].

A local population health survey has reported that 41.1% of persons between the ages of 45 and 64 are at medium-to-high risk of developing cardiovascular diseases over the next 10 years [6]. Most of the cardiometabolic diseases are attributable to health behaviours. An international study identified risk factors for coronary heart disease and validated the non-laboratory INTERHEART Risk Score (IHRS), which is mainly calculated based on behavioural risk factors, including smoking, stress and physical activity [7]. Also, another study among 32 countries in Asia, Africa, Australia, Europe, the Middle East and USA reported that over 90% of the population attributable risks of stroke could be explained by behavioural risk factors measured by IHRS [8]. Proactive measures to moderate these modifiable risk factors are crucial to halt the increasing trend of cardiometabolic disease.

Health coaching interventions are generally effective for managing chronic diseases, including cancer, heart disease, diabetes and hypertension [9]. A systematic review reported health coaching significantly increased physical activity, improved physical and mental health status in patients with chronic disease [10]. Health coaching interventions assist patients to participate actively in their health care, and health coaches collaborate with patients by giving support and promoting self-efficacy in disease management [11]. Despite the widespread use of evidence based health coaching in chronic disease management and prevention of complication, there is fewer attention on the effects of health coaching in primary disease prevention.

Therefore, a large-scale, robust clinical trial examining the effects of health coaching in reducing the cardiometabolic risk in middle-aged adults is warranted. The purpose of this study is to address the research gap by evaluating the effects of health coaching programme on increasing health promoting behaviours in middle-aged adults with cardiometabolic risk.

ELIGIBILITY:
Inclusion Criteria:

* aged 40-64 years;
* have a non-laboratory INTERHEART risk score (IHRS) of 10 or higher;
* can communicate in Cantonese;
* able to give informed consent.

Exclusion Criteria:

* previous diagnosis of transient ischemic attack, stroke, myocardial infarction, atrial fibrillation, coronary heart disease, heart failure, dementia and chronic renal failure;
* currently on medication to control hyperlipidemia, diabetes or hypertension;
* with eye or retinal disease;
* diagnosis of terminal disease with an expected life expectancy less than 12 months;
* currently participating in any other clinical trial;
* currently participating in any other structured lifestyle-based or exercise-based programme.

Ages: 40 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 202 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2023-03-01 (Estimated); Study Completion 2023-03-01 (Estimated)

PRIMARY OUTCOMES:
Change in health promoting behaviours | Change from baseline at 3 months and 6 months post allocation
  The Chinese version of Health Promoting Lifestyle Profile II (HPLP II) , including health responsibility (9 items), nutrition (9 items), physical activity (8 items) and stress management (8 items), measure the practice of health-promoting behaviours

SECONDARY OUTCOMES:
Change in cardiometabolic risk | Change from baseline at 3 months and 6 months post allocation
  Non-laboratory INTERHEART Risk Score (IHRS) assess the risk of cardiometabolic disease
Change in stroke risk | Change from baseline at 3 months and 6 months post allocation
  Automatic retinal image analysis (ARIA)-stroke will be used to quantify stroke risk
Change in self-efficacy of adopting health promoting behaviours | Change from baseline at 3 months and 6 months post allocation
  Adapted version of the Diabetes Mellitus Type II Self Efficacy Scale will be used to rate the participants level of confidence in various behaviours
Change in psychological distress | Change from baseline at 3 months and 6 months post allocation
  The Chinese version of the shorter version of Depression Anxiety Stress Scales (DASS) developed by Lovibond and Lovibond in 1995 will be used
Change in sleep quality | Change from baseline at 3 months and 6 months post allocation
  The Chinese version of the Pittsburg Sleep Quality Index developed by Buysse and team in 1988 will be used
Change in physical activities | Change from baseline at 3 months and 6 months post allocation
  International Physical Activity Questionnaire - Chinese (IPAQ-C), a short version, 9-item scale, will be used to assess the level of physical activities
Change in systolic blood pressure | Change from baseline at 3 months and 6 months post allocation
  Blood pressure measurement using an electronic sphygmomanometer
Change in diastolic blood pressure | Change from baseline at 3 months and 6 months post allocation
  Blood pressure measurement using an electronic sphygmomanometer
Change in Body Mass Index | Change from baseline at 3 months and 6 months post allocation
  Body Mass Index will be calculated by the measured height and weight
Change in waist-hip-ratio | Change from baseline at 3 months and 6 months post allocation
  Waist-hip-ration will be calculated by the measured waist and hip circumference
Change in blood glucose | Change from baseline at 3 months and 6 months post allocation
  Point of care testing of blood for glucose
Change in blood total cholesterol | Change from baseline at 3 months and 6 months post allocation
  Point of care testing of blood for total cholesterol
Change in blood urate | Change from baseline at 3 months and 6 months post allocation
  Point of care testing of blood for urate

CONTACTS AND LOCATIONS:
Overall Officials: Zoe Kwok, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- The Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhang D, Tang X, Shen P, Si Y, Liu X, Xu Z, Wu J, Zhang J, Lu P, Lin H, Gao P. Multimorbidity of cardiometabolic diseases: prevalence and risk for mortality from one million Chinese adults in a longitudinal cohort study. BMJ Open. 2019 Mar 3;9(3):e024476. doi: 10.1136/bmjopen-2018-024476. PMID 30833320
- [Background] 2. Centre of Health Protection. Death rates by leading causes of death, 2001-2019. Hong Kong SAR government: 2020.
- [Background] Guo F, Moellering DR, Garvey WT. The progression of cardiometabolic disease: validation of a new cardiometabolic disease staging system applicable to obesity. Obesity (Silver Spring). 2014 Jan;22(1):110-8. doi: 10.1002/oby.20585. Epub 2013 Sep 5. PMID 23894121
- [Background] GBD 2019 Diseases and Injuries Collaborators. Global burden of 369 diseases and injuries in 204 countries and territories, 1990-2019: a systematic analysis for the Global Burden of Disease Study 2019. Lancet. 2020 Oct 17;396(10258):1204-1222. doi: 10.1016/S0140-6736(20)30925-9. PMID 33069326
- [Background] Kaffashian S, Dugravot A, Brunner EJ, Sabia S, Ankri J, Kivimaki M, Singh-Manoux A. Midlife stroke risk and cognitive decline: a 10-year follow-up of the Whitehall II cohort study. Alzheimers Dement. 2013 Sep;9(5):572-9. doi: 10.1016/j.jalz.2012.07.001. Epub 2012 Nov 28. PMID 23199495
- [Background] 6. Centre for Health Protection. Population Health Survey 2014/2015. Hong Kong SAR Government.: 2017.
- [Background] McGorrian C, Yusuf S, Islam S, Jung H, Rangarajan S, Avezum A, Prabhakaran D, Almahmeed W, Rumboldt Z, Budaj A, Dans AL, Gerstein HC, Teo K, Anand SS; INTERHEART Investigators. Estimating modifiable coronary heart disease risk in multiple regions of the world: the INTERHEART Modifiable Risk Score. Eur Heart J. 2011 Mar;32(5):581-9. doi: 10.1093/eurheartj/ehq448. Epub 2010 Dec 22. PMID 21177699
- [Background] O'Donnell MJ, Chin SL, Rangarajan S, Xavier D, Liu L, Zhang H, Rao-Melacini P, Zhang X, Pais P, Agapay S, Lopez-Jaramillo P, Damasceno A, Langhorne P, McQueen MJ, Rosengren A, Dehghan M, Hankey GJ, Dans AL, Elsayed A, Avezum A, Mondo C, Diener HC, Ryglewicz D, Czlonkowska A, Pogosova N, Weimar C, Iqbal R, Diaz R, Yusoff K, Yusufali A, Oguz A, Wang X, Penaherrera E, Lanas F, Ogah OS, Ogunniyi A, Iversen HK, Malaga G, Rumboldt Z, Oveisgharan S, Al Hussain F, Magazi D, Nilanont Y, Ferguson J, Pare G, Yusuf S; INTERSTROKE investigators. Global and regional effects of potentially modifiable risk factors associated with acute stroke in 32 countries (INTERSTROKE): a case-control study. Lancet. 2016 Aug 20;388(10046):761-75. doi: 10.1016/S0140-6736(16)30506-2. Epub 2016 Jul 16. PMID 27431356
- [Background] Wolever RQ, Simmons LA, Sforzo GA, Dill D, Kaye M, Bechard EM, Southard ME, Kennedy M, Vosloo J, Yang N. A Systematic Review of the Literature on Health and Wellness Coaching: Defining a Key Behavioral intervention in Healthcare. Glob Adv Health Med. 2013 Jul;2(4):38-57. doi: 10.7453/gahmj.2013.042. PMID 24416684
- [Background] Kivela K, Elo S, Kyngas H, Kaariainen M. The effects of health coaching on adult patients with chronic diseases: a systematic review. Patient Educ Couns. 2014 Nov;97(2):147-57. doi: 10.1016/j.pec.2014.07.026. Epub 2014 Aug 1. PMID 25127667
- [Background] 11. UCSF Center for Excellence in Primary Care. Health coach curriculum. University of California: 2014.
- [Background] 12. WalkerSN, Hill-PolereckyDM. Psychometric evaluation of the Health-Promoting Lifestyle Profile II. Unpublished manuscript, University of Nebraska Medical Center 1996.
- [Background] Lee RL, Loke AJ. Health-promoting behaviors and psychosocial well-being of university students in Hong Kong. Public Health Nurs. 2005 May-Jun;22(3):209-20. doi: 10.1111/j.0737-1209.2005.220304.x. PMID 15982194
- [Background] 14. ZeeB, LeeJ, LiQ, MokV, KongA, ChiangL, et al. Stroke risk assessment for the community by automatic retinal image analysis using fundus photograph. Qual Prim Care 2016;24:114-24.
- [Background] Brouwer-Goossensen D, van Genugten L, Lingsma HF, Dippel DWJ, Koudstaal PJ, den Hertog HM. Self-efficacy for health-related behaviour change in patients with TIA or minor ischemic stroke. Psychol Health. 2018 Dec;33(12):1490-1501. doi: 10.1080/08870446.2018.1508686. Epub 2018 Dec 30. PMID 30596258
- [Background] 16. CheungAKY, ToriCD, LamCLK. Psychosocial correlates of medically unexplained physical symptoms in primary care settings: a cross-sectional study in Hong Kong. Hong Kong Pract 2012;34:99-105.
- [Background] Tsai PS, Wang SY, Wang MY, Su CT, Yang TT, Huang CJ, Fang SC. Psychometric evaluation of the Chinese version of the Pittsburgh Sleep Quality Index (CPSQI) in primary insomnia and control subjects. Qual Life Res. 2005 Oct;14(8):1943-52. doi: 10.1007/s11136-005-4346-x. PMID 16155782
- [Background] Macfarlane DJ, Lee CC, Ho EY, Chan KL, Chan DT. Reliability and validity of the Chinese version of IPAQ (short, last 7 days). J Sci Med Sport. 2007 Feb;10(1):45-51. doi: 10.1016/j.jsams.2006.05.003. Epub 2006 Jun 30. PMID 16807105